CLINICAL TRIAL: NCT06106438
Title: Pulmonary Function Tests in Children and Adolescents With End Stage Renal Disease On Regular Hemodialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Mahmoud Othman, Assistant Lecturer, Assiut University
Other Study IDs: PFTs in children with ESRD
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: End Stage Renal Disease on Dialysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to study pulmonary function tests in children with ESRD on regular HD and its correlation with dialysis duration and other various risk factors

DETAILED DESCRIPTION:
End stage renal disease (ESRD) is irreversible and progressive disease which characterized by irreversible loss of kidney function. The ESRD is terminal and final pathway that resulted eventually in most of the patients suffering from medical problems affecting their renal function. Patients with ESRD need renal replacement therapy once they are established the ESRD stage via and that may either be achieved by dialysis (hemodialysis or peritoneal dialysis) or need kidney transplantation so as to be able to keep functioning normal renal life. There was an observed increase in the morbidity and mortality in ESRD patients because of the presence of the renal replacement therapy (HD or renal transplantation). Despite that ESRD may appear as a single organ dysfunction, it also affects multiple organs with variable and numerous complications which resulted in multi-organ dysfunction so the systemic complications presented in ESRD patients are very important .

One of the most important of these complications is the respiratory system dysfunction related to renal dysfunction which is a very common complication in ESRD patients . Rising in the blood urea level, may be the cause that affects the respiratory system in the form of pulmonary edema, pleural effusion and acute respiratory distress syndrome (ARDS) .

Dialysis may have beneficial effects at least in the initial stages of some respiratory disorders among CKD patients without primary lung disease. It may lead to improvement of respiratory symptoms and even pulmonary function test values.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents(more than seven years old and less than 18 years old) with ESRD on regular maintenance HD for at least six months before inclusion on the study

Exclusion Criteria:

* patients with age less than seven years or more than 18
* patients with congenital heart diseases
* patient with bronchial asthma
* patient with musculoskeletal disorders
* patient who were unable to cooperate

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents(more than seven years old and less than 18 years old) with ESRD on regular maintenance HD for at least six months before inclusion on the study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary function tests | one year from january 2024 to december 2024
  by spirometry including The forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC), peak expiratory flow (PEF), and FEV1/FVC ratio and forced expiratory flow (FEF) Pulmonary function tests will be measured before and after hemodialysis session

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mahrous El Tellawy, Professor, Study Chair — Assiut University

REFERENCES:
- [Background] Bush A, Gabriel R. Pulmonary function in chronic renal failure: effects of dialysis and transplantation. Thorax. 1991 Jun;46(6):424-8. doi: 10.1136/thx.46.6.424. PMID 1858080
- [Background] Navari K, Farshidi H, Pour-Reza-Gholi F, Nafar M, Zand S, Sohrab Pour H, Eqbal Eftekhaari T. Spirometry parameters in patients undergoing hemodialysis with bicarbonate and acetate dialysates. Iran J Kidney Dis. 2008 Jul;2(3):149-53. PMID 19377229
- [Background] Senatore M, Buemi M, Di Somma A, Sapio C, Gallo GC. [Respiratory function abnormalities in uremic patients]. G Ital Nefrol. 2004 Jan-Feb;21(1):29-33. Italian. PMID 15356844
- See also: Spirometric Parameters: Hemodialysis Compared to Peritoneal Dialysis — https://jctm.mums.ac.ir/article_4376.html